CLINICAL TRIAL: NCT01741818
Title: The Cutoff Point for Caval Index and Its Correlation With Central Venous Pressure and Plasma Lactate Level for Assessing Patients in Hypovolemic Hemorrhagic States
Status: Completed | Type: Observational
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Keihan Golshani, Assistant Professor of Emergency Medicine, Isfahan University of Medical Sciences
Other Study IDs: IUMS-14746
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: IVC Collapsibility Index; Hemorrhagic Shock
Keywords: IVC; ultrasonography; IVC collapsibility index; IVC diameter
MeSH Terms: conditions — Shock, Hemorrhagic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group B: CVP less than 8cmH2o
  Interventions: Other: Measuring IVC collapsibility index by bedside ultrasonography

INTERVENTIONS:
Other: Measuring IVC collapsibility index by bedside ultrasonography

SUMMARY:
The purpose of this study is to determine the cutoff point for IVC collapsibility index (by Bedside Ultrasonographic technique) for cases in hypovolemic hemorrhagic shock with CVP measures less than 8 cmH2o.

ELIGIBILITY:
Inclusion Criteria:

* Hypovolemic hemorrhagic subjects (class II or more)if they were more than 18 years old and CVC insertion was indicated for them.

Exclusion Criteria:

* a history of Renal failure, Congestive Heart Failure, use of negative inotropic agents, presence of any contraindication for CVC insertion or failed ones and inability for measuring IVC by bUS were considered for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cases in hypovolemic hemorrhagic status (class II or more) that presented to our ED
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
IVC collapsibility index | within the first 5 minutes

SECONDARY OUTCOMES:
Serum lactate level | within the first 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Keihan Golshani, MD., Study Chair — Isfahan University of Medical Sciences
Locations (2):
- Iran (2):
  - Emergency Department of alzahra General Hospital, Isfahan University of Medical Sciences, Isfahan, Isfahan
  - Kerman University of Medical Sciences, Kerman, Kerman